CLINICAL TRIAL: NCT02203071
Title: Comparison of BioCartilage Versus Marrow Stimulating Procedure for Cartilage Defects of the Knee
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, James Stannard, Principal Investigator, University of Missouri-Columbia
Other Study IDs: 1211220
Record Dates: First submitted 2014-06-19; First posted 2014-07-29 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Defect of Articular Cartilage
Keywords: sports; injury; knee; pain; cartilage
MeSH Terms: conditions — Wounds and Injuries; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MSP with BioCartilage: Patients receiving marrow stimulating procedure with BioCartilage adjunct.
- MSP without BioCartilage: Patients receiving marrow stimulating procedure without BioCartilage.

SUMMARY:
Subjects will be selected among the investigators' patient population who are already scheduled to receive a marrow stimulating procedure (MSP), with or without the addition of BioCartilage.

During the surgical operation for MSP, a portion of the patient's blood is taken out and used to form a patch to cover a cartilage defect of the knee. Currently it is considered standard of care to either form the patch using only a portion of the patient's blood, or form the patch using a portion of the patient's blood combined with an FDA-approved augmentation such as BioCartilage.

This study will collect outcomes data and MRI for patients that are undergoing MSP with and without BioCartilage augmentation, then compare the data between those who received BioCartilage and those who did not.

The primary endpoint is to determine whether subjects receiving a marrow stimulating procedure (MSP) augmented with BioCartilage have improved outcomes (measured using quality of life indicators, functional outcomes, and MRI) compared to subjects who receive MSP without the use of BioCartilage.

DETAILED DESCRIPTION:
Recent developments in the treatment of articular cartilage defects have resulted in several techniques that involve the stimulation of native cellular components for the purpose of differentiation and proliferation in the cartilage defect. Techniques of interest for this study are the use of microfracture combined with platelet rich plasma (PRP), and a recently developed augmentation of the microfracture procedure-BioCartilage.

The microfracture procedure is performed with PowerPick. During the procedure, a patient with focal cartilage defect undergoes arthroscopic debridement of the defect before microfracture is used to create holes in the subchondral plate in order to provide access to mesenchymal stem cells (MSCs). To complete this marrow stimulating procedure (MSP), the microfractured region is filled with PRP harvested intraoperatively from the patient. A fibrin glue is then used to cover the defect and hold the PRP repair in place.

This basic MSP has been shown to regenerate cartilage tissue and improve joint function. Microfracture treatments using PRP are "shown to have good to excellent short-term outcomes in appropriately indicated patients" (Abrams, Mall, Fortier, Roller, & Cole, 2013), however successful long-term outcomes have not been demonstrated in the literature.

BioCartilage, a novel therapy developed by Arthrex Inc, is implemented as an augmentation of the basic approach of using microfracture and PRP. All aspects of the procedure, as well as indications for the procedure, are the same as the basic MSP described above, except the PRP is combined with BioCartilage powder, which acts as a scaffolding for cellular growth. BioCartilage is an FDA approved augmentation of microfracture treatment with PRP, and the powder itself contains no living cells.

Animal models using BioCartilage have provided data that supports the assertion that the BioCartilage augmentation may improve outcomes for patients who receive it; however there is currently no published human clinical outcomes data available for using BioCartilage (Abrams et al., 2013).

ELIGIBILITY:
Inclusion Criteria:

I. Inclusion in the study will be considered when all of the following conditions are met:

* The subject is a candidate for the use of a MSP with microfracture and PRP, with or without augmentation with BioCartilage, for treatment of a focal defect of the knee (trochlea or femoral condyle).
* The subject is 18-years of age or greater
* The subject is able and willing to consent to participate in the study
* The subject is expected to be able to safely undergo MRI at the 1-year follow-up visit (no contraindications present, such as metal implants)
* Infection or inflammatory arthropathy (such as rheumatoid arthritis) is absent in the operative knee

Exclusion Criteria:

II. Exclusion from the study will be determined by any one of the following conditions being met:

* The subject is undergoing bilateral knee surgery
* The subject is unwilling, or unable to consent due to psychiatric condition or legal incompetence
* The subject is either pregnant, or a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from Missouri Orthopaedic Institute's patient population.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P Stannard, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Missouri Orthopaedic Institute, Columbia, Missouri, United States

REFERENCES:
- [Derived] Shah SS, Lee S, Mithoefer K. Next-Generation Marrow Stimulation Technology for Cartilage Repair: Basic Science to Clinical Application. JBJS Rev. 2021 Jan 19;9(1):e20.00090. doi: 10.2106/JBJS.RVW.20.00090. PMID 33512974

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 Subjects were intra-operative screen failures.
Period: Overall Study
Arm/Group | MSP With BioCartilage | MSP Without BioCartilage
Started | 13 | 6
Completed | 10 | 5
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Population: There are six subjects who failed to meet intra-operative criteria for study participation.
Groups:
- Total: Total of all reporting groups
Arm/Group | MSP Without BioCartilage | MSP With BioCartilage | Total
Number analyzed (Participants) | 6 | 13 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 12 | 18
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 1 | 7 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 13 | 19
BMI (Body Mass Index) [Mean (Full Range); unit: kg/m^2] | 31.2 [29 to 34] | 30.6 [22 to 32] | 30.8 [22 to 34]

OUTCOME MEASURES:

1. Primary Outcome: MRI Repair Tissue Comparison
Description: The primary endpoint is to determine whether subjects receiving a marrow stimulating procedure (MSP) augmented with BioCartilage have improved outcomes (MRI) compared to subjects who receive MSP without the use of BioCartilage. Quantitative (%fill) and qualitative (tissue quality) MRI assessments of repair tissue will be performed by a musculoskeletal (MSK) radiologist who is blinded to treatment group, and compared for differences between treatment groups.
Time Frame: 1 year post-operatively
Population: There were 6 screen fails and 10 enrolled subjects who did not complete the study. Fifteen patients who were screened, consented, and enrolled, completed the 2-year study. Five patients who completed the study were assigned to the MSP treatment group and ten were assigned to the BioCartilage treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | MSP With BioCartilage | MSP Without BioCartilage
Number analyzed (Participants) | 13 | 6
Participants
  >50% fill, isointense | 10 | 2
  <50% fill, non-isointense | 3 | 4
Statistical Analysis 1: Comparison: MSP With BioCartilage vs MSP Without BioCartilage; Test type: Superiority; p = 0.61, Fisher Exact

2. Secondary Outcome: Short Form-12 Health Survey (SF-12)
Description: The 12-item Short Form Survey (SF-12) is a general health questionnaire. The SF-12 was constructed using questions drawn from each of the 8 dimensions of the MOS 36 item Short Form Survey (SF-36). It is designed to have similar performance to the SF-36, while taking less time to complete. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Approximately 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MSP With BioCartilage | MSP Without BioCartilage
Number analyzed (Participants) | 10 | 5
score on a scale
  Physical Health Composite Scores | 51.4 (7) | 43.4 (10)
  Mental Health Composite Scores | 56.1 (7) | 59.2 (4.3)
Statistical Analysis 1: Comparison: MSP With BioCartilage vs MSP Without BioCartilage; Test type: Superiority; p = .001, t-test, 2 sided

3. Other Pre Specified Outcome: Marx Activity Rating Scale
Description: The Marx Scale consists of four questions concerning four activities or actions: running, cutting, deceleration, and pivoting. The patient or survey respondent is asked to report on the frequency with which they performed the activity in their healthiest state within the past year. The four knee functions are rated on a 5-point scale of frequency and scores are added up to a minimum score of 0 and a maximum of 16 points, with a higher score indicating more frequent participation.
Time Frame: Approximately 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MSP With BioCartilage | MSP Without BioCartilage
Number analyzed (Participants) | 10 | 5
score on a scale | 9.5 (5) | 3.4 (4.2)
Statistical Analysis 1: Comparison: MSP With BioCartilage vs MSP Without BioCartilage; Test type: Superiority; p > 0.11, t-test, 2 sided

4. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcomes Score (KOOS)
Description: The Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Time Frame: Approximately 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MSP With BioCartilage | MSP Without BioCartilage
Number analyzed (Participants) | 10 | 5
score on a scale | 85.9 (12) | 71.6 (18)
Statistical Analysis 1: Comparison: MSP With BioCartilage vs MSP Without BioCartilage; Test type: Superiority; p < 0.007, ANOVA

5. Other Pre Specified Outcome: International Knee Documentation Committee (IKDC) Subjective Portion
Description: The IKDC Questionnaire is a subjective scale that provides patients with an overall function score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee. Meanwhile, the sports activity subscale focuses on functions like going up and down the stairs, rising from a chair, squatting and jumping. The knee function subscale asks patients one simple question: how is their knee at present versus how was their knee prior to injury?
  Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
Time Frame: Approximately 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MSP With BioCartilage | MSP Without BioCartilage
Number analyzed (Participants) | 10 | 5
score on a scale | 76.7 (13.3) | 68.9 (22.8)
Statistical Analysis 1: Comparison: MSP With BioCartilage vs MSP Without BioCartilage; Test type: Superiority; p < 0.001, ANOVA

6. Other Pre Specified Outcome: Number of Participants Who Were Able To Return To Return to Work or Sports Activity
Description: This is a two question survey administered to subjects that obtains subjective data "Yes / No" regarding whether the subject has been able to return to work or sports activity since surgery.
Time Frame: Approximately 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MSP With BioCartilage | MSP Without BioCartilage
Number analyzed (Participants) | 10 | 5
Participants | 9 | 4
Statistical Analysis 1: Comparison: MSP With BioCartilage vs MSP Without BioCartilage; Test type: Superiority; p = 1, Fisher Exact

ADVERSE EVENTS:
Time Frame: The time period for collection of adverse events is 2 years post intervention.
Arm/Group | MSP With BioCartilage | MSP Without BioCartilage
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/71/NCT02203071/Prot_SAP_000.pdf